CLINICAL TRIAL: NCT05640830
Title: A Phase 1B/2 Study of Trastuzumab, Bevacizumab with Paclitaxel for HER2-positive Gastric Cancer in a Second-line Therapy (TREAZURE)
Brief Title: Trastuzumab, Bevacizumab with Paclitaxel for HER2-positive Gastric Cancer in a Second-line Therapy
Acronym: TREAZURE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hoe Koo, Principal Investigator, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREAZURE
Record Dates: First submitted 2022-11-25; First posted 2022-12-07 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: HER2-positive Advanced Gastric Cancer
Keywords: HER2-positive gastric cancer; trastuzumab, bevacizumab & paclitaxel
MeSH Terms: interventions — Trastuzumab; Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TREAZURE (Experimental): This is a single arm study. Trastuzumab has been administered at 6 mg/kg every 3 weeks after initial loading of 8 mg/kg during the first anticancer treatment, so in the second anticancer treatment, 4 mg/kg is administered every 2 weeks to maintain the same concentration. Bevacizumab is administered at 5 mg/kg at 2-weekly intervals used in metastatic colorectal cancer. Paclitaxel is administered on a standard schedule of 80 mg/m2 for 3 consecutive weeks followed by a 1-week break as an existing weekly regimen, and when side effects occur, the weekly dose is reduced by 25% to 60 mg/m2 for 3 weeks or administered every 2 weeks. Administer 80 mg/m2. Administration of this drug is set as one cycle of 4 weeks.
  Interventions: Drug: trastuzumab, bevacizumab with paclitaxel (triple combination)

INTERVENTIONS:
Drug: trastuzumab, bevacizumab with paclitaxel (triple combination) — Trastuzumab 4 mg/kg Day 1, 15 Bevacizumab 5 mg/kg Day 1, 15 Paclitaxel 80 mg/m2 Day 1, 8, 15 every 4 weeks

SUMMARY:
This is a multicenter, open-label, prospective, phase 2 study of trastuzumab, bevacizumab, and paclitaxel as second-line treatment for patients with HER2-positive advanced gastric cancer who had progressed on first-line chemotherapy including trastuzumab or anti-HER2 agents.

DETAILED DESCRIPTION:
Trastuzumab has been administered at 6 mg/kg every 3 weeks after initial loading of 8 mg/kg during the first anticancer treatment, so in the second anticancer treatment, 4 mg/kg is administered every 2 weeks to maintain the same concentration. Bevacizumab is administered at 5 mg/kg at 2-weekly intervals used in metastatic colorectal cancer. Paclitaxel is administered on a standard schedule of 80 mg/m2 for 3 consecutive weeks followed by a 1-week break as an existing weekly regimen, and when side effects occur, the weekly dose is reduced by 25% to 60 mg/m2 for 3 weeks or administered every 2 weeks. Administer 80 mg/m2. Administration of this drug is set as one cycle of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HER2-positive advanced gastric cancer

   * Defined as IHC 2+, which is IHC 3+ or SISH + (or FISH) evaluated by laboratory tests. (SISH positivity is defined as the ratio of the HER2 gene copy number to the CEP17 signal ≥ 2.0)
   * or significant overexpression of HER2 protein on target proteomic analysis (multiple reaction monitoring)
2. Patients who have progressed in response to one systemic anticancer therapy for advanced gastric cancer
3. Patients who are willing and able to write a written consent form for this trial.
4. Patients aged 19 years or older at the time of signing the subject consent form.
5. Patients with measurable or evaluable lesions according to RECIST 1.1.
6. ECOG activity status 0, 1 or 2
7. as patients with adequate organ function

   * Absolute neutrophil (ANC) ≥1.0 x 109/L, platelet ≥100 x 109/L, hemoglobin ≥9 g/dL, serum creatinine ≤1.5 x ULN, total bilirubin ≤3.0 mg on laboratory tests within 2 weeks before starting treatment /dL, AST/ALT ≤5 x ULN
   * Echocardiogram EF ≥55% or MUGA scan ≥50%

Exclusion Criteria:

1. Patients who have received chemotherapy, radiation therapy, immunotherapy or targeted therapy for gastric cancer within the past 2 weeks.
2. Patients who have experienced Grade 3-4 gastrointestinal bleeding within 3 months
3. Patients who have experienced an arteriovascular embolism event, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular disorder, or unstable angina within 6 months
4. Ongoing or active infection, symptomatic congestive heart failure, unstable angina, symptomatic or poorly controlled cardiac arrhythmias, uncontrolled thrombotic or hemorrhagic disorders, or any other serious medical disorder not controlled in the investigator's judgment patient with
5. Patients with a history of gastrointestinal perforation or fistula within 6 months.
6. Concomitant diagnosis of cancer in another site or history of active malignant tumor within the past 3 years

   * Excluding fully cured basal cell carcinoma and thyroid cancer, in situ cervical cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 36 months
  Defined as the time from the start of treatment to the date of documented disease progression (according to RECIST 1.1) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hoe Koo, MD,PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yonemura Y, Ninomiya I, Yamaguchi A, Fushida S, Kimura H, Ohoyama S, Miyazaki I, Endou Y, Tanaka M, Sasaki T. Evaluation of immunoreactivity for erbB-2 protein as a marker of poor short term prognosis in gastric cancer. Cancer Res. 1991 Feb 1;51(3):1034-8. PMID 1670998
- [Background] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Background] Guideline Committee of the Korean Gastric Cancer Association (KGCA), Development Working Group & Review Panel. Korean Practice Guideline for Gastric Cancer 2018: an Evidence-based, Multi-disciplinary Approach. J Gastric Cancer. 2019 Mar;19(1):1-48. doi: 10.5230/jgc.2019.19.e8. Epub 2019 Mar 19. No abstract available. PMID 30944757
- [Background] Shitara K, Bang YJ, Iwasa S, Sugimoto N, Ryu MH, Sakai D, Chung HC, Kawakami H, Yabusaki H, Lee J, Saito K, Kawaguchi Y, Kamio T, Kojima A, Sugihara M, Yamaguchi K; DESTINY-Gastric01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Gastric Cancer. N Engl J Med. 2020 Jun 18;382(25):2419-2430. doi: 10.1056/NEJMoa2004413. Epub 2020 May 29. PMID 32469182
- [Background] du Manoir JM, Francia G, Man S, Mossoba M, Medin JA, Viloria-Petit A, Hicklin DJ, Emmenegger U, Kerbel RS. Strategies for delaying or treating in vivo acquired resistance to trastuzumab in human breast cancer xenografts. Clin Cancer Res. 2006 Feb 1;12(3 Pt 1):904-16. doi: 10.1158/1078-0432.CCR-05-1109. PMID 16467105
- [Background] Singh R, Kim WJ, Kim PH, Hong HJ. Combined blockade of HER2 and VEGF exerts greater growth inhibition of HER2-overexpressing gastric cancer xenografts than individual blockade. Exp Mol Med. 2013 Nov 1;45(11):e52. doi: 10.1038/emm.2013.111. PMID 24176949
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Background] Meulendijks D, Beerepoot LV, Boot H, de Groot JW, Los M, Boers JE, Vanhoutvin SA, Polee MB, Beeker A, Portielje JE, de Jong RS, Goey SH, Kuiper M, Sikorska K, Beijnen JH, Tesselaar ME, Schellens JH, Cats A. Trastuzumab and bevacizumab combined with docetaxel, oxaliplatin and capecitabine as first-line treatment of advanced HER2-positive gastric cancer: a multicenter phase II study. Invest New Drugs. 2016 Feb;34(1):119-28. doi: 10.1007/s10637-015-0309-4. Epub 2015 Dec 8. PMID 26643663
- [Background] Jung M, Ryu MH, Oh DY, Kang M, Zang DY, Hwang IG, Lee KW, Kim KH, Shim BY, Song EK, Sym SJ, Han HS, Park YL, Kim JS, Lee HW, Lee MH, Koo DH, Song HS, Lee N, Yang SH, Choi DR, Hong YS, Lee KE, Maeng CH, Baek JH, Kim S, Kim YH, Rha SY, Cho JY, Kang YK. Efficacy and tolerability of ramucirumab monotherapy or in combination with paclitaxel in gastric cancer patients from the Expanded Access Program Cohort by the Korean Cancer Study Group (KCSG). Gastric Cancer. 2018 Sep;21(5):819-830. doi: 10.1007/s10120-018-0806-1. Epub 2018 Feb 9. PMID 29427038
- [Background] Mun DG, Bhin J, Kim S, Kim H, Jung JH, Jung Y, Jang YE, Park JM, Kim H, Jung Y, Lee H, Bae J, Back S, Kim SJ, Kim J, Park H, Li H, Hwang KB, Park YS, Yook JH, Kim BS, Kwon SY, Ryu SW, Park DY, Jeon TY, Kim DH, Lee JH, Han SU, Song KS, Park D, Park JW, Rodriguez H, Kim J, Lee H, Kim KP, Yang EG, Kim HK, Paek E, Lee S, Lee SW, Hwang D. Proteogenomic Characterization of Human Early-Onset Gastric Cancer. Cancer Cell. 2019 Jan 14;35(1):111-124.e10. doi: 10.1016/j.ccell.2018.12.003. PMID 30645970